CLINICAL TRIAL: NCT01058395
Title: Phase I Study of Minocycline in a Dose Escalation Study as a Safe, Efficacious Therapeutic Intervention for Moderate and Severe TBI in Humans
Brief Title: Safety and Feasibility of Minocycline in the Treatment of Traumatic Brain Injury (TBI)
Acronym: TBI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Jay M Meythaler, MD, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #H133A080044 -01; IND# 104298 (Registry Identifier: FDA)
Record Dates: First submitted 2010-01-19; First posted 2010-01-28 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Minocycline; Outcome
MeSH Terms: conditions — Brain Injuries, Traumatic; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 800 mg loading then 200 mg Q12 (Experimental): Minocycline 800 mg. loading followed by 200 mg. Q 12 hours.
  Interventions: Drug: Minocycline
- 800 mg loading then 400 mg Q12 (Experimental): Minocycline 800 mg. loading followed by 400 mg. Q 12 hours.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 800 mg loading followed by 200 mg Q12 or Minocycline 800 mg loading followed by 400 mg Q12 will be delivered in an open-label study for seven days intravenously in one of two different dosing tiers to assess safety and toxicity per FDA recommendations. There will be tow different arms or groups differing by the amount of minocycline given over 7 days.
  Other Names: Minocin

SUMMARY:
The purpose of this study is:

1. To assess the safety and feasibility of minocycline administration after TBI in a dose escalation study at two different doses over 7 days.
2. To assess the pharmacokinetic characteristics of two different dosing regimens of minocycline in TBI patients, the effect on biochemical markers of neuroprotective mechanisms, and effect on neurobehavioral and functional outcome.
3. To begin initial assessment of the efficacy of minocycline as a therapeutic agent for severe human TBI.

DETAILED DESCRIPTION:
The purpose of this preliminary study is to test the hypothesis that administration of minocycline to humans with moderate and severe TBI is both safe and feasible in the acute post-injury setting, and to characterize its disposition and effects on biomarkers of traumatic CNS injury in a Phase IIa trial. The data collected will serve as the basis for a larger Phase IIb clinical trial in a randomized placebo-controlled parallel group design, to investigate further its potential safety and efficacy as a therapeutic agent for severe human TBI.

Tetracycline derivatives, including doxycycline and minocycline, have been shown to be neuroprotective when given after traumatic brain injury (TBI) and ischemia in rodents. In particular, reduced lesion volume and improved neurological outcome have been demonstrated following minocycline treatment of TBI. The proposed mechanism for these observations is multifactorial, and includes inhibition of microglial activation, caspase-mediated apoptosis, and the excitotoxic N-methyl-D-aspartic acid (NMDA) pathway. Because comparable inflammatory, excitotoxic and apoptotic pathways have also been implicated in human TBI, we hypothesize that administration of minocycline will confer neuroprotection after moderate to severe TBI in that milieu as well, with the potential for significant clinical benefit. Minocycline is highly lipophilic, and thus penetrates the human central nervous system (CNS). In addition, it has been shown to be safe when used in non-traumatic human neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male , 18 to 75 years of age, irrespective of race;
* Ability to provide written informed consent or have legal representative provide written informed consent;
* Must be enrolled in the study within 6 of injury and meet the following criteria:

  * GCS score of 12 or less within the first 4 hours of injury;
  * Evidence of neurological injury on computer tomography (CT) of the head;
  * No known allergy to minocycline or other contraindication to receiving this medication.
* Presence of central venous catheter;
* Participants must not have a known life-threatening disease prior to the brain injury: However, individuals with a stable medical illness in the opinion of the investigator may be allowed to enter the study;
* Participants are not to be on any other interventional studies aimed at enhancing neurorecovery;
* Participants are not to be receiving immunosuppressant agents prior to study enrollment.

Exclusion Criteria:

* Participant is a female;
* Participants, guardians or legal representatives who are unwilling to cooperate with the investigation;
* Participants who have received any other investigational drug within 30 days of injury;
* Participants known to have severe ischemic heart disease or congestive heart failure, myocardial infarction, spinal cord injury with ongoing deficits, cancer or any other severe illnesses that in the opinion of the investigator would affect the assessment of therapy;
* Participants with an ongoing neurological disease/condition or previous stroke or TBI;
* Known clinical sequelae of spinal cord injury;
* Massive cerebral hemisphere or brainstem hematoma, incompatible with survival;
* History of major depression requiring the use of the medication at the time of injury;
* Multiple trauma which in the opinion of the investigator, would jeopardize the assessment of therapy;
* Participants who have any type of penetrating head injury;
* Participants receiving chronic steroid treatment;
* Participants receiving isotretinoin;
* Lack of informed consent signed by either the participant or the subject's legal representative;
* Prior TBI, brain tumor, cerebral vascular event, or other stable brain insult;
* Prior history of Pseudotumor cerebri ;
* Patients with known renal failure, BUN/ Creatinine 20:1; creatinine > 2 mg/dl;
* Patients with known hepatic failure, AST/ALT> 3 x Upper Limit of Normal;
* Thrombocytopenia < 75,000/mm;
* Known allergy or sensitivity to any of the tetracyclines or any of the components of the product formulation.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay M Meythaler, MD, Principal Investigator — Wayne State University; Kristina Freese, PA, Study Director — Wayne State University Dept. PM&R Oakwood; John Fath, MD, Principal Investigator — Oakwood Hospital Dearborn, Trauma Surgery Director; Allen Lamb, DO, Study Director — Oakwood Southshore Hospital
Locations (2):
- United States (2):
  - Oakwood Dearborn Hospital, Dearborn, Michigan
  - Oakwood Southshore Hospital, Trenton, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meythaler J, Fath J, Fuerst D, Zokary H, Freese K, Martin HB, Reineke J, Peduzzi-Nelson J, Roskos PT. Safety and feasibility of minocycline in treatment of acute traumatic brain injury. Brain Inj. 2019;33(5):679-689. doi: 10.1080/02699052.2019.1566968. Epub 2019 Feb 12. PMID 30744442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 800 mg Loading Then 200 mg Q12 | 800 mg Loading Then 400 mg Q12
Started | 7 | 8
Completed | 4 (Two died, and one was lost to followup.) | 7 (One died after enrollment. The patient died in the first 48 hours.)
Not Completed | 3 | 1
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 800 mg Loading Then 200 mg Q12 | 800 mg Loading Then 400 mg Q12 | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 13
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 46 [21 to 71] | 40 [21 to 64] | 43 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Disability Rating Scale
  Participants
    United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Disability Rating Scale
Description: The main outcome measure after the safety data was the Disability Rating Scale (DRS). It is a 29 point scale with 29 being a severe vegetative state. It is reliable across time and demonstrates better sensitivity than the Glasgow Outcome Scale.It has been a standard primary outcome measure for most pharmaceutical studies for TBI, and was required by the FDA for the IND approval.
Time Frame: 4 weeks and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 800 mg Loading Then 200 mg Q12 | 800 mg Loading Then 400 mg Q12
Number analyzed (Participants) | 4 | 7
units on a scale
  DRS at 4 weeks | 12.5 (7.7) | 9.7 (6.9)
  DRS at 3 months | 8.5 (9.9) | 6.0 (6.1)
Statistical Analysis 1: Comparison: 800 mg Loading Then 200 mg Q12 vs 800 mg Loading Then 400 mg Q12; DRS levels changes at from 4 weeks to 3 months comparing the different doses; Test type: Superiority — Comparison between groups at 3 months (primary). Comparison between the 2 tiers; p = 0.021, ANCOVA — P-value; Threshold for significance was P-value < 0.05
Statistical Analysis 2: Comparison: 800 mg Loading Then 200 mg Q12 vs 800 mg Loading Then 400 mg Q12; Null hypothesis is that there is no difference between groups in the DRS scores at 3 months; Test type: Superiority; p = 0.258, t-test, 2 sided
Statistical Analysis 3: Comparison: 800 mg Loading Then 200 mg Q12 vs 800 mg Loading Then 400 mg Q12; Null hypothesis is that there is no difference between groups in the DRS scores at 4 weeks; Test type: Superiority — t-test; p = 0.541, t-test, 2 sided

2. Secondary Outcome: Drug Levels
Description: Serum samples were collected for assessment of minocycline concentrations at the estimated time of steady-state concentrations. Serum concentrations were assessed on Day 4. Data reported will be pKa levels 2 hours after AM dose.
Time Frame: 4 days after start
Population: Those we were able to obtain levels on reliably and could run against standards. This only turned out to be the first tier level. Descriptive data only
Measure: Mean (Full Range); unit: mcg/ml
Arm/Group | 800 mg Loading Then 200 mg Q12
Number analyzed (Participants) | 4
mcg/ml | 21.7 [6.2 to 61.3]

3. Post Hoc Outcome: Aspartate Aminotransferase (AST) Levels
Description: AST levels measured daily from day 1 to day 7 evaluated by ANOVA. Mean values on day 7 reported for the two tiers.
  Elevations may indicate Liver dysfunction due to medication.
Time Frame: day 1 change to day 7 day, ANOVA, mean value on day 7 reported
Population: Levels are compared for the two tiers
Measure: Mean (Full Range); unit: U/L
Arm/Group | 800 mg Loading Then 200 mg Q12 | 800 mg Loading Then 400 mg Q12
Number analyzed (Participants) | 4 | 7
U/L | 88.0 [31 to 245] | 264 [30 to 1092]
Statistical Analysis 1: Comparison: 800 mg Loading Then 200 mg Q12 vs 800 mg Loading Then 400 mg Q12; Test type: Superiority; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 176

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious Adverse l event medical or laboratory related to the use of the medication.
Arm/Group | 800 mg Loading Then 200 mg Q12 | 800 mg Loading Then 400 mg Q12
All-Cause Mortality (participants affected / at risk) | 2/7 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 800 mg Loading Then 200 mg Q12 (N=7) | 800 mg Loading Then 400 mg Q12 (N=8)
Medical (Nervous system disorders) | 7 | 8

LIMITATIONS AND CAVEATS:
Preliminary open label study, generally to assess the safety of the use of Minocycline at the dosages specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes